CLINICAL TRIAL: NCT00330239
Title: Paroxetine Treatment in Outpatients With Comorbid PTSD and Substance Dependence
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CPMS-857
Record Dates: First submitted 2006-05-25; First posted 2006-05-26 (Estimated); Last update posted 2007-10-03 (Estimated); Status verified 2007-10

CONDITIONS: PTSD
Keywords: Substance Abuse; Trauma; Dependence
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Substance-Related Disorders; Wounds and Injuries

INTERVENTIONS:
Drug: Paroxetine CR

SUMMARY:
Pharmacotherapy has demonstrated efficacy in a number of controlled trials in the treatment of PTSD. The selective serotonin reuptake inhibitors have proven particularly useful in treating this disorder. Currently there are two selective serotonin reuptake inhibitors (Zoloft® and Paxil®), that have been FDA approved for treating PTSD. Coincidentally, this same class of medications has also been shown to have efficacy in some trials in decreasing alcohol consumption in heavy drinkers. The goal of the proposed study is to preliminarily investigate the efficacy of Paxil® (paroxetine), in decreasing symptoms of PTSD as well as decreasing substance use, in individuals with concurrent substance dependence and PTSD. The type of paroxetine used in this trial will be Paxil CR®, which is a sustained release formulation of paroxetine, which has fewer side effects and greater tolerability. This is a particularly important issue in substance using populations because medication compliance is generally poor.

Two specific hypotheses will be tested. 1) Individuals who receive Paxil CR® will have a greater improvement in their PTSD symptoms (based on CAPS-2 and CGI) than those who receive placebo. 2) Individuals who receive Paxil CR® will have greater improvement in their substance use outcomes (based on UDS and TLFB) than will those who receive placebo.

DETAILED DESCRIPTION:
Participants who meet all inclusion and no exclusion criteria will be randomized with a 1:1 ratio to receive either Paxil CR or placebo for 12 weeks. Medication will be initiated at 12.5mg/day and will be increased weekly as tolerated to a maximum dose of 50mg/day. Participants will be seen weekly and will be assessed for side effects, substance use since last visit, urine drug screen, breathalyzer readings, vital signs and symptoms of PTSD (TOP-8)at each visit. The Davidson Trauma Scale will be completed every two weeks, and the CAPS-2 and MADRS will be completed monthly. Those who complete the first 12 weeks of double-blind study medication will be eligible to receive open label medication for an additional 12 weeks. Medication will be initiated at 12.5mg and increased every 3 days as tolerated to the terminal dose in the double-blind phase, then adjusted as needed. Participants will come in for assessments every two weeks of the open-label phase. Blood will be drawn for blood chemistries and hematology at screening and weeks 12 and 24. Urine pregnancy tests will be performed for women of childbearing potential at baseline and again at weeks 4, 12 and 24.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 65
* Outpatients who meet DSM-IV criteria for PTSD, chronic subtype, based on CAPS-1
* Must have a minimum score of 50 on the CAPS-2 at Baseline
* Must meet DSM-IV criteria for a substance dependence disorder in the last 3 months (excluding caffeine and nicotine)
* Must be able to read English
* Must give written informed consent

Exclusion Criteria:

* Individuals with a primary psychiatric disorder other than PTSD
* Individuals with an uncontrolled neurologic condition that could confound the results of the study (e.g. seizure disorder)
* Individuals with an uncontrolled medical condition that may adversely affect the conduct of this trial or jeopardize subject safety
* Concomitant use of other psychotropic medications (intermittent use of diphenhydramine and zolpidem will be allowed during the study) see concommitant meds on page 5 of the protocol
* Women of childbearing potential who are pregnant, lactating or refuse to use adequate forms of birth control
* Individuals who have failed an adequate trial of paroxetine in the past
* Current suicidal or homicidal risk
* Currently receiving trauma-specific psychotherapy
* Individuals taking any herbal psychoactive treatments (e.g. St. John's Wart)
* Individuals engaged in compensation litigation whereby personal gain would be achieved from prolonged symptoms of PTSD or any other psychiatric disorder
* Individuals, who in the investigator's opinion would be unable to comply with study procedures or assessments

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2003-01; Study Completion 2005-05

PRIMARY OUTCOMES:
Clinician Administered PTSD Scale (CAPS)
Clinical Global Impressions Scale

SECONDARY OUTCOMES:
Davidson Trauma Scale
Time-Line Follow-Back

CONTACTS AND LOCATIONS:
Overall Officials: Susan C Sonne, PharmD, Principal Investigator — Medical University of South Carolina; Kathleen T Brady, MD, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States